CLINICAL TRIAL: NCT05758727
Title: The Efficacy of Home-based Strength and Tai-chi Exercise Snacking for Improving Physical Function in Taiwanese and British Older Adults: a Randomised Control Trial.
Brief Title: Homebased Strength and Tai-chi Exercise Snacking for Improving Physical Function in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Ian-Ju Liang, Doctoral student, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EP 20/21 082
Record Dates: First submitted 2023-02-15; First posted 2023-03-07 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Older Adults
Keywords: Exercise snacking; Tai-chi snacking; Older adults; Homebased exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based exercise group (Experimental): This group will be asked to practise the 'exercise snacking and Tai-chi snacking' exercises once each and record the exercise bouts in a log book.
  Interventions: Other: Exercise intervention
- Control group (No Intervention): Usual care control group

INTERVENTIONS:
Other: Exercise intervention — The exercise programme is progressive and has three levels. Each bout of exercise and Tai-chi snacking consists of 5 exercises. Each exercise is performed for one minute with one minute rest in between. For exercise snacking movements (including leg exercise, shoulder exercise, single leg exercise, arm exercise, and ankle exercise), participants are encouraged to complete as many repetitions as possible of that exercise in that minute. For Tai-chi snacking movements (including single leg squat, trunk rotation, single leg stand, hip and knee exercise, and ankle mobility exercise), participants are encouraged to complete repetitions of each exercise at a self-selected pace that is comfortable for them to maintain for the full minute, with the aim being to complete the movements as accurately and smoothly as possible (based on correct posture and proper alignment).
  Arms: Home-based exercise group

SUMMARY:
Engaging in muscle strength and balance (S&B) exercises and has numerous health benefits for older adults, promoting greater mobility, reducing risk of falling, and overall improved health and wellbeing. Given the rising age of global populations, reducing the burden associated with lost physical function is essential to minimise health and social care costs. Unfortunately, very few older adults engage in sufficient S&B exercise to reap these benefits, with a lack of time, self-efficacy and access to leisure facilities cited as the key barriers. Finding innovative ways promote an acceptable and engaging format of S&B exercise is consequently a public health priority.

One novel way that aims to address typical barriers to participation in older adults is through the promotion of exercise 'snacks', as opposed to a more traditional, lengthy structured exercise session at a leisure centre. Exercise snacking describes short bursts of exercise that are designed to be undertaken over a short period in the home environment and without the need for any specialised exercise clothing or equipment. In the initial laboratory and cross-sectional and pilot intervention research, the investigators have been testing two formats of 5-minute, twice-daily, strength exercise- and tai-chi-snacking, which has been shown to be acceptable and feasible to implement in older adults. This protocol presents initial efficacy for evoking improved physical function in people aged 65 years or more. The investigators' remote study demonstrated that remote assessment and delivery of 4-week exercise and tai-chi snacking interventions were acceptable and feasible. However, qualitative feedback indicated that exercise programmes may be more acceptable and interesting with simpler tai-chi movements and exercise snacking programme with upper body movements. Nevertheless, the investigators only recruited healthy older adults, doing short-term interventions in previous studies. This study aims to test the effectiveness of progressive S&B interventions over a sustained period in pre-frail older adults.

DETAILED DESCRIPTION:
This study will take place over approximately 3 months and involve 5 assessments remotely. A subset of 60 participants will be assessed in person to validate the remote assessment and undergo more in-depth assessments.

Assessment 1: Familiarisation Participants will be directed to a web page with the participant information sheet and a consent tick box. Participants will then complete an online screening questionnaire that will assess eligibility. After this, participants will undertake a familiarisation session either online (all participants) or in person (lab participants only) to become accustomed to the physical function tests and undergo an exercise safety assessment.

Assessment 2: Baseline assessment. After familiarisation, eligible participants will then complete an online baseline questionnaire assessing demographic details, physical activity levels and psychological outcomes. A functional assessment will be arranged over video calling software, and in the laboratory for the lab participants. Functional outcomes will be completed at this visit. Following the baseline assessment participants will be randomised to either the intervention group, or the waitlist control group.

Assessment 3 and 4: Mid intervention. Participants in the intervention group will be given an exercise teaching video and written instructions on how to safely perform the exercise at home by email. The intervention will take place over 12 weeks and consists of three progressive phases that will be self-selected by participants. The participants will be asked to do the exercises and progress to the next level if they pass the progress criteria which will be clearly explained in the exercise guides and instructional videos. The participants will also be asked to record self-reported exercise logs and RPE for each session they complete. Participants will undergo follow-up assessments at weeks 4 and 8 through video calls and in person (if in the lab study).

Assessment 5: Follow-up assessment. After 12 weeks, participants will complete another online survey containing all psychosocial variables and an evaluation of the usefulness and acceptability of their assigned exercise activities. Participants will also undergo follow-up physical performance tests through video calls and in person (if in the lab study) and a subset will undergo a qualitative evaluation to provide further feedback on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* People aged 65 or greater and are able to perform daily physical activity independently.
* Not regularly engaging in recreational sports or structured exercise (once a week or more).
* Citizen of UK or Taiwan.
* Individuals who are able to do the 5 reps sit-to-stand in less than 60s and the feet side-by-side stand for at least 10s, following the initial safety screening.

Exclusion Criteria:

* Individuals with current ongoing medication or treatment for injuries or illness that would impact on any of the study outcomes.
* Individuals with a current musculoskeletal injury that would preclude participation in exercise ascertained through preliminary screening.
* Individuals with contraindications to exercise including chest pain, dizziness, or loss of consciousness, or who have been instructed by their doctor to only do physical activity recommended by them.
* Individuals who have been diagnosed with dementia.
* Individuals who are unable to consent for themselves or complete the familiarisation / baseline screening by themselves.
* Individuals who score more than 8 on the Short Physical Performance Battery, score more than 6 between strength and balance sections, or score zero on any component of the test.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Changes of Short Physical Performance Battery (SPPB) between every 4 weeks | 12-weeks (week 0, week 4, week 8, week 12)
  Participants will be asked to do the SPPB test which includes balance test, gait speed test, and chair stand test.

SECONDARY OUTCOMES:
1RM of leg press | 12-weeks (week 0, week 4, week 8, week 12)
  Participants will be asked to perform leg press on Keiser leg press machine.
Balance function | 12-weeks (week 0, week 4, week 8, week 12)
  Single-leg stand
Strength function | 12-weeks (week 0, week 4, week 8, week 12)
  60 second sit-to-stand test
Agility function | 12-weeks (week 0, week 4, week 8, week 12)
  Timed-up-and-go
Flexibility | 12-weeks (week 0, week 4, week 8, week 12)
  Chair sit and reach test
Quality of life and wellbeing: Life Satisfaction Scale | 12-weeks (week 0, week 4, week 8, week 12)
  A 5-item scale designed to measure global cognitive judgments of one's life satisfaction which uses a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. Individuals score 31-35 are classified as 'Extremely Satisfied', 26-30 as 'Satisfied', 21-25 as 'Slightly satisfied', 20 as 'Neutral', 15-19 as 'Slightly dissatisfied', 10-14 as 'Dissatisfied', and 5-9 as 'Extremely Dissatisfied'.
Physical activity level: the instrumental activities of daily living (IADL) | 12-weeks (week 0, week 4, week 8, week 12)
  An 8-topic instrument to determine older adults' capability of living independently. Each topic is given a score of 0 or 1. A person is judged adequate to live independently if scored 1 and is judged to need assistant if scored 0.
Physical activity level: the International Physical Activity Questionnaire for elderly (IPAQ-E) (short form) | 12-weeks (week 0, week 4, week 8, week 12)
  The short version of the IPAQ-E assesses physical activity in older adults using different domains including sedentary activities, walking (light-intensity activities), moderate-intensity activities and vigorous intensity activities. Participants are asked to provide the time and frequency they spend doing different-intensity activities in the last 7 days by the day of questionnaire completion. IPAQ data are calculated and presented into metabolic equivalent of task (MET).
Current mental health: Subjective Vitality Index | 12-weeks (week 0, week 4, week 8, week 12)
  The Subjective Vitality Scale is a 7-item self-report instrument to measure one's level of vitality. The score is calculated by assigning scores of 1-7 to the response categories from "not at all true," "somewhat true," to "very true,", and then adding together the scores for the seven questions. The total score for the seven items ranges from 0 to 21. The higher the participants scored, the better vitality the participants had.
Self-confidence for exercise: Self-Efficacy for Exercise (SEE) Scale | 12-weeks (week 0, week 4, week 8, week 12)
  This scale is a 9-item self-report of exercise self-efficacy. Total score is calculated by summing the responses to each question, assigning scores of 1-10 to the response categories from "not confident," to "very confident,". This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Self-confidence for exercise: Perceived Competence for Exercise Scale | 12-weeks (week 0, week 4, week 8, week 12)
  This scale is a 4-item self-report of exercise self-efficacy. Total score is calculated by summing the responses to each question, assigning scores of 1-7 to the response categories from "not at all true," "somewhat true," to "very true,". This scale has a range of total scores from 0-28. A higher score indicates higher self-efficacy for exercise.
Attitudes to exercise: Multidimensional Outcome Expectations for Exercise Scale (MOEES) | 12-weeks (week 0, week 4, week 8, week 12)
  This scale is a 15-item self-report of one's beliefs or expectations about the benefits of regular exercise or physical activity. Total score is calculated by summing the responses to each question, assigning scores of 1-5 to the response categories from "strongly disagree," "neutral," to "strongly agree,". A higher score indicates greater positive attitudes to exercise.
Attitudes to exercise: the Self-Report Habit Index | 12-weeks (week 0, week 4, week 8, week 12)
  This scale is a 12-item self-report of one's beliefs about the benefits of exercise. Total score is calculated by summing the responses to each question, assigning scores of 1-7 to the response categories from "not at all true," "somewhat true," to "very true,". A higher score indicates greater positive attitudes to exercise.
Acceptability of the intervention: Theoretical framework of acceptability questionnaire | 12-weeks (week 4, week 8, week 12)
  Acceptability was measured with an 8-item questionnaire based on the dimensions of the theoretical framework of acceptability (TFA). Total score is calculated by summing the responses to each question, assigning scores of 1-5 to the response categories from "completely unacceptable," "no opinion," to "completely acceptable,". A higher score indicates greater acceptability to the exercise programme.
General health: Short Form Health Survey (SF-36) | 12-weeks (week 0, week 4, week 8, week 12)
  The SF-36 is a multi-purpose survey designed to capture participants perceptions of their own health and well-being. The SF-36 has 36 items grouped in 8 dimensions: physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health. It includes combinations of 5-point scales, 3-point scales, and dichotomous (yes/no) items. The instrument's scores are norm-based: a score of 50 = average. A higher score indicates greater health condition ones have.
Mental health and wellbeing: the Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS) | 12-weeks (week 0, week 4, week 8, week 12)
  A 14-item scale with subjective wellbeing and psychological functioning questions for assessing mental health. The score is calculated by assigning scores of 1-5 to the response categories from "none of the time," "some of the time," to "all of the time,", and then adding together the scores for the 14 questions. The total score ranges from 14 to 70. The higher the participants scored, the better wellbeing the participants had.
Quality of life: EQ-5D-5L | 12-weeks (week 0, week 4, week 8, week 12)
  EQ-5D-5L has 5 dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and one subjective EQ VAS score, which is a 0-100 scale where participants were asked to score their overall health on the day of questionnaire completion. regarding the 5 dimensions, the score is assessed by assigning scores of levels 1-5 to the response indicates from no problem, slight to moderate problems, to severe problems, and unable to/extreme problems.
Attitudes to exercise: the Behaviour Regulation Exercise Questionnaire (BREQ-3) | 12-weeks (week 0, week 4, week 8, week 12)
  A 24-item self-report of one's attitudes toward exercise underlying self-determination theory. It indicates amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, and intrinsic regulation toward exercise, using 4-point scales from 0-4 to the response categories from "not true for me," to "very true for me,". The higher the score ones get, the more positive attitudes for exercise ones have.

CONTACTS AND LOCATIONS:
Overall Officials: Max Western, Study Chair — Department for Health, University of Bath
Locations (1):
- Department for Health, University of Bath, Bath, Bath And North East Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No